CLINICAL TRIAL: NCT03500315
Title: HOPE in Action Prospective Multicenter, Clinical Trial of Deceased HIVD+ Kidney Transplants for HIV+ Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00141138; U01AI134591 (NIH)
Record Dates: First submitted 2018-04-02; First posted 2018-04-18 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIV D+/R+ (Experimental): HIV-infected individuals that accept an organ from an HIV-infected deceased donor - enrollment 100
  Interventions: Other: HIV D+/R+
- HIV D-/R+ (No Intervention): HIV-infected individuals that accept an organ from an HIV-uninfected deceased donor -enrollment 100
- HIV D-/R+ (observational) (No Intervention): HIV-infected individuals that accept an organ from an HIV-uninfected deceased donor and randomized to observational group - enrollment 200

INTERVENTIONS:
Other: HIV D+/R+ — Kidney from an HIV-infected deceased donor
  Arms: HIV D+/R+

SUMMARY:
The primary objective of this study is to determine if an HIV-infected deceased kidney donor (HIVD+) transplant is safe with regards to major transplant-related and HIV-related complications.

DETAILED DESCRIPTION:
This study will evaluate if receiving a kidney transplant from an HIV-infected deceased kidney donor is safe with regards to survival and major transplant-related and HIV-related complications compared to receiving a kidney from an HIV-uninfected deceased kidney donor (HIVD-). Those participants who have accepted an HIVD- organ will be randomized to be followed in the full study or followed in the nested observational group.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets the standard criteria for kidney transplant at the local center.
* Participant is able to understand and provide informed consent.
* Participant meets with an independent advocate per the HIV Organ Policy Equity (HOPE) Act Safeguards.
* Documented HIV infection (by any licensed assay, or documented history of detectable HIV-1 RNA).
* Participant is ≥18 years old.
* Opportunistic complications: if prior history of an opportunistic infection, the participant has received appropriate therapy and has no evidence of active disease.
* Cluster of Differentiation 4 (CD4)+ T-cell: ≥200/µL within 16 weeks of transplant.
* HIV-1 is below 50 copies RNA/mL. Viral blips between 50-400 copies allowed as long as there are not consecutive measurements >200 copies/mL.
* Participant is willing to comply with all medication related to their transplant and HIV management.
* For participant with a history of aspergillus colonization or disease, no evidence of active disease.
* The participant must have, or be willing to start seeing, a primary medical care provider with expertise in HIV management.
* All participants participating in sexual activity that could lead to pregnancy must use an FDA approved method of birth control.
* Participant is not suffering from significant wasting (e.g. body mass index <21) thought to be related to HIV disease.

Exclusion Criteria:

* Participant has a history of progressive multifocal leukoencephalopathy (PML) or primary central nervous system (CNS) lymphoma.
* Participant is pregnant or breastfeeding.
* Past or current medical problems or findings from medical history, physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks or may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Composite event, time to first death or graft failure or serious adverse event (SAE) or HIV breakthrough or opportunistic infection | From date of transplant through administrative censorship at study completion, up to 4 years
  Time to first of any of the following events: death or graft failure or serious adverse event (SAE) or HIV breakthrough or HIV virologic failure or opportunistic infection

SECONDARY OUTCOMES:
Pre-transplant mortality | From date of enrollment to date of transplant or death of any cause, whichever comes first, assessed up to 4 years
  Time to mortality while enrolled before transplant (survival framework)
Graft failure | From date of transplant through administrative censorship at study completion, up to 4 years
  Time to mortality or re-transplant or return to maintenance dialysis (survival framework)
Rate of serious adverse events | From date of transplant through graft failure or administrative censorship at study completion, up to year 4
  Count of post-transplant serious adverse events per person-year as assessed by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0
6-month acute rejection | From date of transplant to end of month 6
  Proportion of recipients who experience acute rejection as measured by biopsy using Banff 2015 criteria: Borderline changes: 'Suspicious' for acute T-cell mediated rejection.This category is used when no intimal arteritis is present, but there are foci of mild tubulitis (t1, t2, or t3) with minor interstitial infiltration (i0 or i1) or interstitial infiltration (i2, i3) with mild (t1) tubulitis. Acute T-cell mediated rejection:Grade from IA defined as cases with significant interstitial infiltration (>25% of parenchyma affected, i2 or i3) and foci of moderate tubulitis (t2) to III defined as cases with 'transmural' arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation (v3)
1-year acute rejection | From date of transplant to end of year 1
  Proportion of recipients who experience acute rejection as measured by biopsy using Banff 2015 criteria: Borderline changes: 'Suspicious' for acute T-cell mediated rejection.This category is used when no intimal arteritis is present, but there are foci of mild tubulitis (t1, t2, or t3) with minor interstitial infiltration (i0 or i1) or interstitial infiltration (i2, i3) with mild (t1) tubulitis. Acute T-cell mediated rejection:Grade from IA defined as cases with significant interstitial infiltration (>25% of parenchyma affected, i2 or i3) and foci of moderate tubulitis (t2) to III defined as cases with 'transmural' arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation (v3)
Incidence of graft rejection | From date of transplant through administrative censorship, up to 4 years
  Cumulative incidence of acute rejection (survival framework) as measured by biopsy using Banff 2015 criteria: Borderline changes: 'Suspicious' for acute T-cell mediated rejection.This category is used when no intimal arteritis is present, but there are foci of mild tubulitis (t1, t2, or t3) with minor interstitial infiltration (i0 or i1) or interstitial infiltration (i2, i3) with mild (t1) tubulitis. Acute T-cell mediated rejection:Grade from IA defined as cases with significant interstitial infiltration (>25% of parenchyma affected, i2 or i3) and foci of moderate tubulitis (t2) to III defined as cases with 'transmural' arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation (v3)
Graft function - Proportion eGFR <60 mL/min/1.73 m2 | 3 months post-transplant
  Proportion of transplant recipients with glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) < 60 mL/min/1.73 m2
Graft function - Proportion eGFR <60 mL/min/1.73 m2 | 6 months post-transplant
  Proportion of transplant recipients with glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) < 60 mL/min/1.73 m2
Graft function - Proportion eGFR <60 mL/min/1.73 m2 | 9 months post-transplant
  Proportion of transplant recipients with glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) < 60 mL/min/1.73 m2
Graft function - Proportion eGFR <60 mL/min/1.73 m2 | 1 year post-transplant
  Proportion of transplant recipients with glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) < 60 mL/min/1.73 m2
Graft function - Proportion eGFR <60 mL/min/1.73 m2 | 2 years post-transplant
  Proportion of participants with glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) < 60 mL/min/1.73 m2
Graft function - Proportion eGFR <60 mL/min/1.73 m2 | 3 years post-transplant
  Proportion of participants with glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) < 60 mL/min/1.73 m2
Graft function -mean eGFR | 3 months post-transplant
  Mean calculated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Graft function-mean eGFR | 6 months post-transplant
  Mean calculated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Graft function-mean eGFR | 9 months post-transplant
  Mean calculated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Graft function-mean eGFR | 1 year post-transplant
  Mean calculated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Graft function-mean eGFR | 2 years post-transplant
  Mean calculated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Graft function-mean eGFR | 3 years post-transplant
  Mean calculated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
Graft function - slope eGFR | From date of transplant to end of follow-up, up to 4 years
  The slope of glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) over time (longitudinal analysis)
Incidence of non-HIV renal disease | 6 months post-transplant
  Cumulative incidence of non HIV-related renal disease as measured by biopsy, e.g. focal segmental glomerulosclerosis
Incidence of non-HIV renal disease | 1 year post-transplant
  Cumulative incidence of non HIV-related renal disease as measured by biopsy, e.g. focal segmental glomerulosclerosis
Incidence of HIV-related renal disease | 6 months post-transplant
  Cumulative incidence of non HIV-related renal disease as measured by biopsy, e.g. HIV-associated nephropathy
Incidence of HIV-related renal disease | 1 year post-transplant
  Cumulative incidence of non HIV-related renal disease as measured by biopsy, e.g. HIV-associated nephropathy
Donor and recipient apolipoprotein L1 (APOL1) | Baseline
  Proportion of transplant recipients with at least 1 apolipoprotein L1 (APOL1) risk variant in donor and recipient
HIV infection of renal allografts | 6 months post-transplant
  Proportion of recipients with HIV seen in laser capture microdissection of renal biopsy
Trajectory of recipient plasma HIV RNA over time | From date of transplant through end of follow-up, up to 4 years
  Analysis of repeated measures of plasma HIV RNA (longitudinal model)
Trajectory of recipient Cluster of Differentiation (CD4) count over time | From date of transplant through end of follow up, up to 4 years
  Analysis of repeated measures of Cluster of Differentiation 4 (CD4) count (longitudinal model)
Incidence of antiretroviral resistance | From date of transplant through end of follow-up, up to 4 years
  Measured by local sites' Clinical Laboratory Improvement Amendments (CLIA) certified lab with episode of HIV breakthrough defined as 2 consecutive plasma HIV viral loads >200 copies/mL or one HIV viral load >1000 copies/mL after a period of virologic control post-transplant
Incidence of X4 tropic virus | From date of transplant through end of follow-up, up to 4 years
  Measured by local sites' Clinical Laboratory Improvement Amendments (CLIA) certified lab with episode of HIV breakthrough defined as 2 consecutive plasma HIV viral loads >200 copies/mL or one HIV viral load >1000 copies/mL after a period of virologic control post-transplant
Incidence of opportunistic infection | From date of transplant through end of follow-up, up to 4 years
  Cumulative incidence of opportunistic infections
Incidence of surgical complications | From date of transplant through year 1
  Number of surgical complications within 1 year of transplant, e.g. delayed closure, wound dehiscence
Incidence of vascular complications | From date of transplant through year 1
  Number of vascular complications within 1 year of transplant
Incidence of viral-related malignancies | From date of transplant through end of follow-up, up to 4 years
  Number of malignancies as determined by local pathology
Incidence of the formation of de novo donor-specific human leukocyte antigen(HLA) antibodies | From date of transplant through end of year 1
  Proportion of participants with a de novo donor-specific HLA antibody as measured and reported by local sites' lab
Composite event, time to first | From date of transplant through end of follow-up, up to 4 years
  Time to first of any of these events: all-cause-mortality or graft failure or renal allograft rejection or HIV breakthrough or HIV virologic failure or AIDS defining illness

CONTACTS AND LOCATIONS:
Overall Officials: Christine Durand, MD, Principal Investigator — Johns Hopkins University
Locations (29):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Georgetown Transplant Institute, Washington D.C., District of Columbia
  - Miami Transplant Institute, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC-University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Methodist Health System Clinical Research Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Durand CM, Massie A, Florman S, Liang T, Rana MM, Friedman-Moraco R, Gilbert A, Stock P, Mehta SA, Mehta S, Stosor V, Pereira MR, Morris MI, Hand J, Aslam S, Malinis M, Haidar G, Small CB, Santos CAQ, Schaenman J, Baddley J, Wojciechowski D, Blumberg EA, Ranganna K, Adebiyi O, Elias N, Castillo-Lugo JA, Giorgakis E, Apewokin S, Brown D, Ostrander D, Eby Y, Desai N, Naqvi F, Bagnasco S, Watson N, Brittain E, Odim J, Redd AD, Tobian AAR, Segev DL; HOPE in Action Investigators. Safety of Kidney Transplantation from Donors with HIV. N Engl J Med. 2024 Oct 17;391(15):1390-1401. doi: 10.1056/NEJMoa2403733. PMID 39413376
- [Derived] Werbel WA, Brown DM, Kusemiju OT, Doby BL, Seaman SM, Redd AD, Eby Y, Fernandez RE, Desai NM, Miller J, Bismut GA, Kirby CS, Schmidt HA, Clarke WA, Seisa M, Petropoulos CJ, Quinn TC, Florman SS, Huprikar S, Rana MM, Friedman-Moraco RJ, Mehta AK, Stock PG, Price JC, Stosor V, Mehta SG, Gilbert AJ, Elias N, Morris MI, Mehta SA, Small CB, Haidar G, Malinis M, Husson JS, Pereira MR, Gupta G, Hand J, Kirchner VA, Agarwal A, Aslam S, Blumberg EA, Wolfe CR, Myer K, Wood RP, Neidlinger N, Strell S, Shuck M, Wilkins H, Wadsworth M, Motter JD, Odim J, Segev DL, Durand CM, Tobian AAR; HOPE in Action Investigators. National Landscape of Human Immunodeficiency Virus-Positive Deceased Organ Donors in the United States. Clin Infect Dis. 2022 Jun 10;74(11):2010-2019. doi: 10.1093/cid/ciab743. PMID 34453519